CLINICAL TRIAL: NCT00378339
Title: Clinical Effects From Implants of Gold Around the Arthrotic Knee Joint. A Randomized, Double Blind, Placebo Controlled Investigation.
Brief Title: Gold Against Pains From Osteoarthrosis in the Knee
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because of lack of approvement from local medical authorities
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ON-04-015-MBL
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Arthritis
Keywords: arthrosis; gold
MeSH Terms: conditions — Arthritis; Osteoarthritis

INTERVENTIONS:
Device: gold berlocks

SUMMARY:
Gold implantation around arthritic joints is a very popular treatment - but the effect has never been controlled.

DETAILED DESCRIPTION:
Randomization between

1. Gold (4 x 3 berlocks, injected under local anesthesia) and
2. Sham operation - only local anesthesia Functional and pain measures reported through the next 6 months.

ELIGIBILITY:
Inclusion Criteria:

Arthrosis in knee joint

Exclusion Criteria:

Need for NSAID

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
VAS

SECONDARY OUTCOMES:
WOMAC

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, Phd, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Frederikshavn, Frederikshavn, Northern Jutland, Denmark